CLINICAL TRIAL: NCT00697229
Title: Study to Evaluate the Immunogenicity and Reactogenicity of GSK Biologicals' MPL-Adjuvanted Recombinant Hepatitis B Vaccine in Comparison With Those of Engerix™-B in Healthy Adult Volunteers Following 2 Different Schedules
Brief Title: Immunogenicity & Reactogenicity of HBV-MPL Vaccine and Engerix™-B in Healthy Adults Following 2 Different Schedules
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Isabelle Harpigny, GSK
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 208129/004
Record Dates: First submitted 2008-06-11; First posted 2008-06-13 (Estimated); Last update posted 2008-06-13 (Estimated); Status verified 2008-06

CONDITIONS: Hepatitis B
Keywords: Hepatitis B; Engerix™-B; Recombinant hepatitis B vaccine
MeSH Terms: conditions — Hepatitis B

ARMS (8):
- Group A (Experimental): Subjects will receive HBV-MPL vaccine in the primary schedule 0, 2 months and will receive a booster dose of HBV-MPL vaccine at 70 months
  Interventions: Biological: HBV-MPL vaccine
- Group B (Experimental): Subjects will receive HBV-MPL vaccine in the primary schedule 0, 2 months and will receive a booster dose of Engerix™-B vaccine at 70 months
  Interventions: Biological: Engerix™-B; Biological: HBV-MPL vaccine
- Group C (Experimental): Subjects will receive Engerix™-B vaccine in the primary schedule 0, 2 months and will receive a booster dose of HBV-MPL vaccine at 70 months
  Interventions: Biological: Engerix™-B
- Group D (Experimental): Subjects will receive Engerix™-B vaccine in the primary schedule 0, 2 months and will receive a booster dose of Engerix™-B vaccine at 70 months
  Interventions: Biological: Engerix™-B; Biological: HBV-MPL vaccine
- Group E (Experimental): Subjects will receive HBV-MPL vaccine in the primary schedule 0, 6 months and will receive a booster dose of HBV-MPL vaccine at 70 months
  Interventions: Biological: HBV-MPL vaccine
- Group F (Experimental): Subjects will receive HBV-MPL vaccine in the primary schedule 0, 6 months and will receive a booster dose of Engerix™-B vaccine at 70 months
  Interventions: Biological: Engerix™-B; Biological: HBV-MPL vaccine
- Group G (Experimental): Subjects will receive Engerix™-B vaccine in the primary schedule 0, 6 months and will receive a booster dose of HBV-MPL vaccine at 70 months
  Interventions: Biological: Engerix™-B
- Group H (Experimental): Subjects will receive Engerix™-B vaccine in the primary schedule 0, 6 months and will receive a booster dose of Engerix™-B vaccine at 70 months
  Interventions: Biological: Engerix™-B; Biological: HBV-MPL vaccine

INTERVENTIONS:
Biological: Engerix™-B — Intramuscular injection, 1 or 3 doses
  Arms: Group B; Group C; Group D; Group F; Group G; Group H
Biological: HBV-MPL vaccine — Intramuscular injection, 1 or 3 doses
  Arms: Group A; Group B; Group D; Group E; Group F; Group H

SUMMARY:
The purpose of this study is to evaluate the safety, immunogenicity and reactogenicity of MPL-adjuvanted recombinant hepatitis B vaccine in comparison with those of Engerix™-B in healthy adult volunteers following two different schedules: 0, 2 months and 0, 6 months

DETAILED DESCRIPTION:
At the time of conduct of this study, the sponsor GlaxoSmithKline was known by its former name SmithKline Beecham

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 40 years old.
* Written informed consent will have been obtained from the subjects.
* Good physical condition as established by physical examination and history taking at the time of entry.
* Female participants will avoid becoming pregnant during the study period and they will have been on a contraceptive program for at least 2 months before entry.

Exclusion Criteria:

* Positive titres for anti hepatitis B antibodies.
* Any vaccination against hepatitis B in the past.
* Elevated serum liver enzymes.
* History of significant and persisting hematologic, hepatic, renal, cardiac or respiratory disease.
* Axillary temperature > 37°C at the time of injection.
* Any acute disease at the moment of entry.
* Chronic alcohol consumption.
* Any chronic drug treatment, including any treatment with immunosuppressive drugs, which in the investigator's opinion, precludes inclusion into the study.
* History of allergic disease likely to be stimulated by any component of the vaccine.
* Administration of any other vaccine(s) or any immunoglobulin during the study period.
* Simultaneous participation in any other clinical trial.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 99 (Actual)
Dates: Start 1992-09; Primary Completion 1996-05 (Actual); Study Completion 1998-12 (Actual)

PRIMARY OUTCOMES:
Anti-hepatitis B surface antigen (HBs) antibody concentrations | One month after the full primary vaccination course and one month after the booster vaccination at 70 months

SECONDARY OUTCOMES:
Anti-HBs antibody concentrations | Months 1, 2, 3, 6, 12, 13, 42
Serious adverse experiences (SAE). | Throughout the study period
Occurrence and intensity of solicited local symptoms | 8-day follow-up after vaccination
Occurrence, intensity and relationship of solicited general symptoms | 8-day follow-up after vaccination
Incidence of unsolicited symptoms | During the 30-day follow-up after vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Clinical Trials Call Center, Wilrijk, Belgium